CLINICAL TRIAL: NCT03975361
Title: Tolerance Checkpoints Upon the B-cell Depletion Plus BAFF Blockade Strategy in Immune Thrombocytopenia (ITP) and Systemic Lupus Erythematosus (SLE) (Checkpoints ITP and SLE)
Brief Title: Autoreactivity Threshold Analysis in Lupus and Immune Thrombocytopenia (Checkpoints ITP and SLE)
Acronym: ITP&SLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP180341; 2019-A00103-54 (Other: IDRCB)
Record Dates: First submitted 2019-05-24; First posted 2019-06-05 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-12

CONDITIONS: Immune Thrombocytopenia (ITP); Systemic Lupus Erythematosus (SLE)
Keywords: Rituximab
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bliss-Believe (Other): Patients included in the BLISS-BELIEVE study (NCT03312907).
  Interventions: Other: Bliss-Believe

INTERVENTIONS:
Other: Bliss-Believe — The samples from the blood samples carried out within the framework of Bliss Believe will be collected for a biological collection. Only one sample of patients included in BLISS BELIEVE STUDY will be obtained during a standard of care visit. It will be 21ml of blood.

SUMMARY:
The aim of this proposal is to test if anti-BAFF antibody can restore a normal threshold of tolerance in patients in two auto-immune diseases along the RITUX-PLUS study in immune thrombocytopenia, and along the Believe study in SLE. This work would help to conclude whether or not the 'double hit' therapy may help to reset the immune system toward a more tolerogenic profile.

The aim is to compare the polyreactivity and autoreactivity, of immature (central tolerance) and naïve B cells (peripheral tolerance) in the peripheral blood along the RITUX-PLUS STUDY and the BLISS BELIEVE study after treatment (B-cell reconstitution time).

ELIGIBILITY:
There are no specific inclusion and exclusion criteria for this study.

The inclusion and exclusion criteria are those of patients enrolled in the RITUX-PLUS (NCT03154385) and BLISS BELIEVE studies (NCT03312907) including the following inclusion criteria:

* individuals are affiliated to social security
* individuals not be placed under judicial protection, guardianship or curatoship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-04-29 (Estimated); Study Completion 2022-04-29 (Estimated)

PRIMARY OUTCOMES:
Number of polyreactive and autoreactive cells in immature and naïve B cells subsets in the peripheral blood | 1 year
  Number of polyreactive and autoreactive cells in immature (central tolerance) and naïve B cells (peripheral tolerance) subsets in the peripheral blood along the RITUX-PLUS and the BLISS BELIEVE studies after treatment (reconstitution time).

CONTACTS AND LOCATIONS:
Overall Officials: Mahevas Matthieu, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Henri Mondor Hospital, Créteil
  - Pitie Salpetriere Hospital, Paris